CLINICAL TRIAL: NCT03196921
Title: A Prospective Cohort to Evaluate the Efficacy and Safety of Oral Encochleated Amphotericin B (CAMB/MAT2203) for the Treatment of Cryptococcal Infection
Brief Title: Efficacy and Safety of Oral Encochleated Amphotericin B for the Treatment of Cryptococcal Infection
Acronym: ORACLE
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Protocol redundancy
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MB-70009
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Cryptococcal Infections
Keywords: amphotericin B; cryptococcal

STUDY DESIGN:
Intervention Model Description: Patients with symptomatic cryptococcal meningitis will be enrolled in treatment arm Patients that are CRAG positive will be enrolled the in prevention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Symptomatic Cryptococcal Meningitis (Experimental): CAMB (Encochleated Amphotericin B)
  Interventions: Drug: Encochleated Amphotericin B
- Asymptomatic Cryptococcal Antigenemia (Experimental): CAMB (Encochleated Amphotericin B)
  Interventions: Drug: Encochleated Amphotericin B

INTERVENTIONS:
Drug: Encochleated Amphotericin B — lipid-crystal nanoparticle formulation of amphotericin B; oral
  Other Names: CAMB; MAT2203

SUMMARY:
This will be an open label phase I/II prospective cohort study to determine the efficacy and safety of CAMB for the treatment and prevention of cryptococcal infection.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection, informed consent, cryptococcal infection present, diagnosed by either: CSF cryptococcal culture, CSF cryptococcal antigen (CRAG), plasma/serum CRAG

Exclusion Criteria:

* Presence of jaundice or known liver cirrhosis, >72 hours antifungal therapy, pregnancy or breastfeeding, unlikely to attend regular clinic visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability of drug over 14 days of dosing | 14-days
  Tolerability of drug as measured by the proportion of doses received versus the number of scheduled doses
Microbiologic clearance of Cryptococcus from the CSF | 14-days

SECONDARY OUTCOMES:
Incidence of adverse events | 14-days
  stratified by symptomatic and asymptomatic subgroups
Survival from cryptococcal infection | 10-weeks
  stratified by symptomatic and asymptomatic subgroups
Pharmacokinetics | 24-hours
  PK parameter of Area Under the Curve (AUC)
Pharmacokinetics | 24-hours
  PK parameter of the maximum concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: David R Boulware, MD, MPH, Principal Investigator — University of Minnesota; Tafese Beyene Tufa, Principal Investigator — Asella Teaching Hospital, Arsi University

IPD SHARING:
Plan to Share IPD: No